CLINICAL TRIAL: NCT03313362
Title: Detecting PNES With Single-channel sEMG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brain Sentinel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PNES-1.5-01.2017
Record Dates: First submitted 2017-10-10; First posted 2017-10-18 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Epilepsy, Motor Partial; Psychogenic Seizures
MeSH Terms: conditions — Epilepsy, Partial, Motor; Psychogenic Nonepileptic Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Subjects admitted to Epilepsy Monitoring Units in the VAMC (Experimental): Subjects being monitored by standard of care, video EEG, in the Epilepsy Monitoring Units in the VAMC will all be placed on a Seizure Monitoring and Alerting System (SPEAC System).
  Interventions: Device: SPEAC System; Device: video EEG

INTERVENTIONS:
Device: SPEAC System — Seizure Monitoring and Alerting System
  Other Names: Brain Sentinel Seizure Monitoring and Alerting System
Device: video EEG — The Video EEG Monitoring Test (VEEG) is a high specialized form of an EEG test in where the patient is continuosly monitored by using a video recorder. This allows doctors to observe brainwaves activity during the time a seizure or spell is occurring.

SUMMARY:
This is a prospective, comparative, multicenter study of subjects being admitted for standard of care therapy in Epilepsy Monitoring Units in the Veteran's Affair (VA) Medical Centers.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a history of suspected epileptic seizures with upper extremity motor involvement, or PNES with upper extremity motor involvement.
2. Is being admitted to a hospital for routine vEEG monitoring related to seizures.
3. Male or Female between the ages 22 to 99.
4. If female and of childbearing potential, has a negative pregnancy test and must not be nursing.
5. Can understand and sign written informed consent, or will have a parent or a legally authorized representative (LAR) who can do so, prior to the performance of any study assessments.
6. Subject and/or Primary Caregiver must be competent to follow all study procedures.
7. Subject/LAR consents to the use of vEEG files, including video/audio recordings, for purposes of this research study.

Exclusion Criteria:

* Intracranial EEG electrodes are being used.

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Test an independent group of epileptologist's ability to classify motor events between epileptic or non-epileptic using sEMG and audio. | 1 year
  To test the null hypothesis that three independent epileptologists categorize, by majority vote, epileptic seizures and psychogenic non-epileptic seizures (identified utilizing vEEG review) correctly in no more than 70% of cases using sEMG and audio. We aim to test the null hypothesis that the epileptologists categorize epileptic seizures and psychogenic non-epileptic seizures correctly in no more than 70% of cases. The observed rate of correct classification will be compared to the rate of 70% under the null hypothesis using a two-sided binomial exact test.

SECONDARY OUTCOMES:
To test the Brain Sentinel® Seizure Monitoring and Alerting System's ability to classify motor events as epileptic or non-epileptic. | 1 Year
  Test the null hypothesis that the Brain Sentinel® Seizure Monitoring and Alerting System categorizes epileptic seizures and psychogenic non-epileptic seizures (identified utilizing vEEG review) correctly in no more than 70% of cases. We aim to test the null hypothesis that the Brain Sentinel® Seizure Monitoring and Alerting System's software categorizes epileptic seizures and psychogenic Nonepileptic seizures correctly in no more than 70% of cases. The observed rate of correct classification will be compared to the rate of 70% under the null hypothesis using a two-sided binomial exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Aatif Husain, MD, Principal Investigator — Epilepsy Center of Excellence (ECoE) at the Durham VA Medical Center in Durham, North Carolina; Alan Towne, MD, Principal Investigator — Epilepsy Center of Excellence (ECoE) at Hunter Holmes McGuire VA Medical Center in Richmond, Virginia; David Chen, MD, Principal Investigator — Epilepsy Center of Excellence (ECoE) at the Michael E. DeBakey VA Medical Center in Houston, Texas
Locations (3):
- United States (3):
  - Durham VAMC, Durham, North Carolina
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia